CLINICAL TRIAL: NCT05181527
Title: Repurposing of Dextromethorphan as an Adjunct Therapy in Patients With Major Depressive Disorder: A Randomized, Group Sequential, Adaptive Design, Controlled Clinical Trial
Brief Title: Repurposing of Dextromethorphan as an Adjunct Therapy in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, RITUPARNA MAITI, Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIIMSBBSR/PGThesis/21-22/74
Record Dates: First submitted 2021-12-16; First posted 2022-01-06 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors; Dextromethorphan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Patients in the control group will get an identical-looking capsule containing placebo (starch) once daily in addition to SSRI.
  Interventions: Drug: Selective Serotonin Reuptake Inhibitors; Drug: Placebo
- Test group (Experimental): Patients in the test group will get Dextromethorphan 30 mg once daily orally as an add-on to ongoing SSRI treatment.
  Interventions: Drug: Selective Serotonin Reuptake Inhibitors; Drug: Dextromethorphan

INTERVENTIONS:
Drug: Selective Serotonin Reuptake Inhibitors — Patients in both the study arms will receive SSRI for 8 weeks.
Drug: Dextromethorphan — Patients in the test group will get Dextromethorphan 30 mg once daily orally as an add-on to ongoing SSRI treatment for 8 weeks.
  Arms: Test group
Drug: Placebo — Patients in the control group will get placebo tablet once daily orally as an add-on to ongoing SSRI treatment for 8 weeks.
  Arms: Control group

SUMMARY:
Therapeutic latency, lack of efficacy, and adverse drug reactions are the major concerns in current antidepressant therapies. One-third of the patients with major depressive disorder do not respond to conventional antidepressants that act through the monoaminergic system. To overcome these treatment hurdles, add-on therapy to standard antidepressant drugs may lead to better therapeutic outcomes. The recent discovery of the rapid and sustained antidepressant effect of subanesthetic dose of ketamine led to many extensive clinical and preclinical research in the recent past and has established the possibilities of NMDA receptors as a potential drug target for depression. As repeated doses of ketamine are related to abusive potential and adverse effects, the search for a similar antidepressant agent with a better safety profile is essential. Dextromethorphan has the property of noncompetitively blocking N-methyl-D-aspartate receptors (like ketamine) with additional serotonin transporter and norepinephrine transporter inhibitory action. So, the investigators expect that adding dextromethorphan to selective serotonin reuptake inhibitors (SSRIs) regimen can improve clinical outcomes in major depressive disorder. The literature search found that to date, there is no randomized controlled trial on Dextromethorphan as add-on therapy to first-line antidepressants like SSRIs. So, the present randomized controlled trial has been planned to evaluate the efficacy and safety of add-on dextromethorphan to SSRIs in major depressive disorder.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common psychiatric disorder with a substantial socioeconomic burden with a global prevalence rate of 16%. The underlying pathophysiology of depression is still not understood completely. Among the different proposed hypotheses, the most accepted is the monoamine hypothesis which is the basis of most of the available drugs like tricyclic antidepressants, Monoamine oxidase Inhibitors, selective serotonin reuptake inhibitors (SSRIs), serotonin and norepinephrine reuptake inhibitors (SNRIs). Although many medications are available, a significant proportion of patients become either non-responders or treatment-resistant depression patients.

Another major concern is the therapeutic lag period with all of these monoaminergic antidepressants. Additionally, most of the available antidepressant drugs have many adverse effects, which increase with increments in dose. The discovery of the rapid and sustained antidepressant effect of subanesthetic dose of ketamine, especially in the treatment of non-responders and treatment-resistant cases leads to many extensive clinical and preclinical research in the recent past. As repeated doses of ketamine are related to abusive potential and many other adverse effects, the search for a similar antidepressant agent is going on, which acts via a similar mechanism with a better safety profile. Dextromethorphan, an FDA-approved over-the-counter antitussive drug, has a similar property of non-competitively blocking N-methyl-D-aspartate receptors of glutamate, like ketamine. Additionally, Dextromethorphan has serotonin transporter inhibitory and NET inhibitory properties, so it can also increase the availability of serotonin in synapses, hence may achieve a synergistic effect with SSRIs. In 2010, US-FDA approved Dextromethorphan plus quinidine (Nuedexta) for use in pseudobulbar affect (PBA), and currently, it is under investigation as a potential antidepressant agent in MDD (NCT01882829, NCT02153502). In the phase, IIa clinical trial by Murrough et al. have reported acceptable tolerability and efficacy of dextromethorphan/quinidine combination in treatment-resistant depression (TRD). Another combination of Dextromethorphan and bupropion is currently in phase III clinical trial for TRD. In the present background, the investigators hypothesize that the major concerns of antidepressant therapy like therapeutic latency, lack of efficacy, and adverse drug reactions may be overcome by adding Dextromethorphan to SSRI in MDD. As SSRIs inhibit CYP2D6, the addition of quinidine with Dextromethorphan may not be reasonable and hence, not considered in the present study. The literature search found that to date, there is no randomized controlled trial on Dextromethorphan as an add-on therapy to first-line antidepressants like SSRIs. So, the present randomized controlled trial has been planned to evaluate the efficacy and safety of add-on dextromethorphan to SSRIs in major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with major depressive disorder of either gender within the age group of 18-65 years
* Patients with MADRS score ≥ 7 and ≤ 34 (patients having mild to moderate MDD).
* Patients who are on a stable dose of Sertraline 50 mg or any other Selective Serotonin Reuptake Inhibitor (SSRI) therapy in equivalent dose for less than equal to 4 weeks.
* Patients who have given written informed consent.

Exclusion Criteria:

* Patients who have been treated with Electro Convulsive Therapy (ECT) recently.
* History of epilepsy, or other major neurological or medical disorders, head trauma.
* Patients with a history of Bipolar Depression (BPD).
* Patients with schizophrenia or other psychotic disorder.
* Patients with suicidal thoughts or risk.
* Patients with cognitive impairment.
* Initiating or stopping formal psychotherapy within six weeks before enrolment.
* Patients with comorbidities like any malignancies, hepatic, renal, cardiovascular,
* neurological or endocrinal, respiratory dysfunction.
* Substance abuse history of psychoactive agents.
* Pregnant and lactating mothers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in severity in depressive symptoms | Baseline and 8 weeks
  Will be assessed by Montgomery-Asberg Depression Rating Scale score. The overall score ranges from 0 to 60. A higher score denotes greater severity of depression.

SECONDARY OUTCOMES:
To evaluate treatment response rate | 8 weeks
  Treatment response rate will be assessed as a percentage of patients showing 50% change in Montgomery-Asberg Depression Rating Scale scores from baseline, after 8-week follow-up.
To evaluate the symptom remission rate | 8 weeks
  Symptom remission rate will be assessed as a percentage of patients achieving Montgomery-Asberg Depression Rating Scale scores <7 at 8-week follow-up.
Severity of depressive symptoms at baseline | At baseline
  Severity of depressive symptoms at baseline will be assessed by Clinical Global Impression- severity (CGI-S) score. The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale and the higher value suggests greater severity of the disease.
To evaluate the improvement in symptoms of depression | 8 weeks
  The improvement in symptoms of depression will be assessed by Clinical Global Impression- Improvement (CGI-I) score. The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale and a lower value suggests greater improvement in symptoms.
To evaluate the neurotrophic effect of the treatment | Baseline and 8 weeks
  The neurotrophic effect of the treatment will be assessed by estimating Serum Brain-Derived Neurotrophic Factor (BDNF) level at baseline and at 8-week.
To evaluate the level of the experimental drug (dextromethorphan) | 8 weeks
  Serum dextromethorphan level will be estimated using high-pressure liquid chromatography (HPLC) at 8 weeks after starting the drug.

CONTACTS AND LOCATIONS:
Overall Officials: Rituparna Maiti, M.D., Principal Investigator — AIIMS, Bhubaneswar
Locations (1):
- All India Institute of Medical Sciences (AIIMS), Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang YT, Wang XL, Feng ST, Chen NH, Wang ZZ, Zhang Y. Novel rapid-acting glutamatergic modulators: Targeting the synaptic plasticity in depression. Pharmacol Res. 2021 Sep;171:105761. doi: 10.1016/j.phrs.2021.105761. Epub 2021 Jul 7. PMID 34242798
- [Result] Lener MS, Kadriu B, Zarate CA Jr. Ketamine and Beyond: Investigations into the Potential of Glutamatergic Agents to Treat Depression. Drugs. 2017 Mar;77(4):381-401. doi: 10.1007/s40265-017-0702-8. PMID 28194724
- [Result] Saavedra JS, Garrett PI, Honeycutt SC, Peterson AM, White JW, Hillhouse TM. Assessment of the rapid and sustained antidepressant-like effects of dextromethorphan in mice. Pharmacol Biochem Behav. 2020 Oct;197:173003. doi: 10.1016/j.pbb.2020.173003. Epub 2020 Aug 2. PMID 32755625
- [Result] Henter ID, Park LT, Zarate CA Jr. Novel Glutamatergic Modulators for the Treatment of Mood Disorders: Current Status. CNS Drugs. 2021 May;35(5):527-543. doi: 10.1007/s40263-021-00816-x. Epub 2021 Apr 26. PMID 33904154
- [Result] Fogaca MV, Wu M, Li C, Li XY, Picciotto MR, Duman RS. Inhibition of GABA interneurons in the mPFC is sufficient and necessary for rapid antidepressant responses. Mol Psychiatry. 2021 Jul;26(7):3277-3291. doi: 10.1038/s41380-020-00916-y. Epub 2020 Oct 17. PMID 33070149
- [Result] Zanos P, Gould TD. Mechanisms of ketamine action as an antidepressant. Mol Psychiatry. 2018 Apr;23(4):801-811. doi: 10.1038/mp.2017.255. Epub 2018 Mar 13. PMID 29532791
- [Result] Nguyen L, Scandinaro AL, Matsumoto RR. Deuterated (d6)-dextromethorphan elicits antidepressant-like effects in mice. Pharmacol Biochem Behav. 2017 Oct;161:30-37. doi: 10.1016/j.pbb.2017.09.005. Epub 2017 Sep 12. PMID 28916283
- [Result] Kamijima K, Kimura M, Kuwahara K, Kitayama Y, Tadori Y. Randomized, double-blind comparison of aripiprazole/sertraline combination and placebo/sertraline combination in patients with major depressive disorder. Psychiatry Clin Neurosci. 2018 Aug;72(8):591-601. doi: 10.1111/pcn.12663. Epub 2018 May 21. PMID 29660207
- [Derived] Maji S, Mishra A, Mohapatra D, Mishra BR, Jena M, Srinivasan A, Maiti R. Early augmentation therapy with dextromethorphan in mild to moderate major depressive disorder: A group sequential, response adaptive randomized controlled trial. Psychiatry Res. 2024 Dec;342:116257. doi: 10.1016/j.psychres.2024.116257. Epub 2024 Nov 8. PMID 39551007
- [Derived] Maji S, Mohapatra D, Jena M, Srinivasan A, Maiti R. Repurposing of dextromethorphan as an adjunct therapy in patients with major depressive disorder: a randomised, group sequential adaptive design, controlled clinical trial protocol. BMJ Open. 2024 Apr 30;14(4):e080500. doi: 10.1136/bmjopen-2023-080500. PMID 38688675